CLINICAL TRIAL: NCT02807701
Title: Comparative Study Between Minimally Invasive Pancreatico-duodenectomy and Open Pancreatico-duodenectomy for Periampullary Tumors
Brief Title: Minimally Invasive Pancreatico-duodenectomy
Acronym: LPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Gastroenterology surgical center, mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPD
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2016-06

CONDITIONS: Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic pancreaticoduodenectomy (Active Comparator): Laparoscopic pancreaticoduodenectomy Under general anesthesia, the patient is placed in a supine position with the legs abducted. Carbon dioxide pneumoperitoneum is established using an open technique through a 10-mm trocar over the umbilicus. A 30 telescope is inserted to examine the peritoneal cavity, liver, stomach, and mesentric vessels.Then 4 to 6 more trocars are inserted under direct vision in the epigastrium and upper quadrants
  1. dissection
  2. reconstruction
  Interventions: Procedure: Laparoscopic pancreaticoduodenectomy
- Open pancreaticoduodenectomy (Active Comparator): Open pancreaticoduodenectomy Abdomen is opened from the Bilateral Subcostal incision. (Chevron's Incision) 2. Abdominal cavity is explored for metastasis especially in liver, base of mesentary, mesocolon and pelvis.
  Dissection Reconstruction Pancreaticogastrostomy Hepaticojejunostomy is next- Done in single layer and can be performed in interrupted or continuous fashion.
  Gastrojejunostomy is the final step of reconstruction.
  Interventions: Procedure: Open pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Laparoscopic pancreaticoduodenectomy — Laparoscopic pancreaticoduodenectomy
  1. dissection
  2. reconstruction
  Other Names: LPD
  Arms: Laparoscopic pancreaticoduodenectomy
Procedure: Open pancreaticoduodenectomy — Open pancreaticoduodenectomy
  Other Names: O PD
  Arms: Open pancreaticoduodenectomy

SUMMARY:
Open pancreaticoduodenectomy (PD) is the standard treatment for a wide array of periampullary and pancreatic diseases including malignant and benign conditions. The outcome of PD has improved over the last two decades due to advances in surgical techniques, anesthesia and perioperative care. Although studies from high volume centers demonstrate reduce in the operative mortality to less than 3%, the postoperative morbidity rate is still ranging from 30% to 60%. Laparoscopic surgery is being used increasingly as a less invasive alternative to traditional interventions for pancreatic resection. Laparoscopic pancreaticoduodenectomy (LPD) is a difficult procedure that has become increasingly popular. Nevertheless, comparative data on outcomes remain limited. In this prospective randomized study, investigators evaluate the safety and feasibility of surgical and oncological outcomes of minimally invasive PD compared to conventional open PD.

DETAILED DESCRIPTION:
Open pancreaticoduodenectomy (PD) is the standard treatment for a wide array of periampullary and pancreatic diseases including malignant and benign conditions. The outcome of PD has improved over the last two decades due to advances in surgical techniques, anesthesia and perioperative care . Although studies from high volume centers demonstrate reduce in the operative mortality to less than 3%, the postoperative morbidity rate is still ranging from 30% to 60%. Laparoscopic surgery is being used increasingly as a less invasive alternative to traditional interventions for pancreatic resection. Laparoscopic pancreaticoduodenectomy (LPD) is a difficult procedure that has become increasingly popular. Nevertheless, comparative data on outcomes remain limited despite several improvements in surgical devices and techniques that have allowed surgeons to approach the pancreas laparoscopically, laparoscopic PD remains challenging. LPD represents one of the most advanced abdominal operations owing to the necessity of a complex dissection and reconstruction. Recent reports note that complete laparoscopic PD including laparoscopic resection and reconstruction is both technically feasible and safe. In this prospective randomized study, investigators evaluate the safety and feasibility of surgical and oncological outcomes of minimally invasive PD compared to conventional open PD

ELIGIBILITY:
Inclusion Criteria:

1. Age from less than 70 years.
2. Tumor size less than or equal 3cm.
3. No vascular invasion.

Exclusion Criteria:

1. Multiple prior abdominal surgeries.
2. Body mass index >40.
3. Locally advanced tumors .
4. Inability to withstand prolonged anesthesia.
5. Tumor size more than 3 cm.
6. Patients who received chemoradiotherapy.
7. Pregnant females.
8. Patients with cirrhotic liver.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
duration of hospital stay | one month
  hospital stay

SECONDARY OUTCOMES:
postoperative pancreatic fistula | 30 days
  Postoperative pancreatic ﬁstula was defined as proposed by the international study group of pancreatic ﬁstula (ISGPF) as any measurable volume of ﬂuid on or after postoperative day (POD) 3 with amylase content greater than 3 times the serum amylase activity, and classified into grades A, B, C .
operative time | intraoperative hours
  total operative time
blood loss | intraoperative hours
  estimated blood loss intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Study Director — Mansoura University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] El Nakeeb A, Salah T, Sultan A, El Hemaly M, Askr W, Ezzat H, Hamdy E, Atef E, El Hanafy E, El-Geidie A, Abdel Wahab M, Abdallah T. Pancreatic anastomotic leakage after pancreaticoduodenectomy. Risk factors, clinical predictors, and management (single center experience). World J Surg. 2013 Jun;37(6):1405-18. doi: 10.1007/s00268-013-1998-5. PMID 23494109
- [Result] El Nakeeb A, Askr W, Mahdy Y, Elgawalby A, El Sorogy M, Abu Zeied M, Abdallah T, Abd Elwahab M. Delayed gastric emptying after pancreaticoduodenectomy. Risk factors, predictors of severity and outcome. A single center experience of 588 cases. J Gastrointest Surg. 2015 Jun;19(6):1093-100. doi: 10.1007/s11605-015-2795-2. Epub 2015 Mar 11. PMID 25759078
- [Result] Senthilnathan P, Srivatsan Gurumurthy S, Gul SI, Sabnis S, Natesan AV, Palanisamy NV, Praveen Raj P, Subbiah R, Ramakrishnan P, Palanivelu C. Long-term results of laparoscopic pancreaticoduodenectomy for pancreatic and periampullary cancer-experience of 130 cases from a tertiary-care center in South India. J Laparoendosc Adv Surg Tech A. 2015 Apr;25(4):295-300. doi: 10.1089/lap.2014.0502. Epub 2015 Mar 19. PMID 25789541
- [Result] Dokmak S, Fteriche FS, Aussilhou B, Bensafta Y, Levy P, Ruszniewski P, Belghiti J, Sauvanet A. Laparoscopic pancreaticoduodenectomy should not be routine for resection of periampullary tumors. J Am Coll Surg. 2015 May;220(5):831-8. doi: 10.1016/j.jamcollsurg.2014.12.052. Epub 2015 Jan 26. PMID 25840531
- [Result] Croome KP, Farnell MB, Que FG, Reid-Lombardo KM, Truty MJ, Nagorney DM, Kendrick ML. Total laparoscopic pancreaticoduodenectomy for pancreatic ductal adenocarcinoma: oncologic advantages over open approaches? Ann Surg. 2014 Oct;260(4):633-8; discussion 638-40. doi: 10.1097/SLA.0000000000000937. PMID 25203880
- [Result] Guerra F, Levi Sandri GB, Amore Bonapasta S, Farsi M, Coratti A. The role of robotics in widening the range of application of minimally invasive surgery for pancreaticoduodenectomy. Pancreatology. 2016 Mar-Apr;16(2):293-4. doi: 10.1016/j.pan.2015.12.007. Epub 2015 Dec 23. No abstract available. PMID 26774496
- See also: mansoura university — http://www.mans.edu.eg/